CLINICAL TRIAL: NCT04237350
Title: Video Screening for Visual Impairment of Infants
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2019-China-7
Record Dates: First submitted 2020-01-14; First posted 2020-01-23 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Behavioral Dynamics; Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- severe visual impairment group: The "severe visual impairment" group is defined as the BCVA of at least one eye outside the 99% referenced range or worse than light perception with structural abnormalities or other examination results.
  Interventions: Behavioral: Video recording for behaviors
- likely healthy group: For the "likely healthy" group, the visual acuity of both eyes is in the 95% referenced range with no structural abnormalities.
  The referenced range could be found in the following publication:
  Mayer, DL., et al. Monocular acuity norms for the Teller Acuity Cards between ages one month and four years. Investigative Ophthalmology & Visual Science. 36(3):671 (1995)
  Interventions: Behavioral: Video recording for behaviors
- mild visual impairment group: The "mild visual impairment" group is defined as the BCVA in the 99% referenced range in both eyes with abnormalities of structure or other examination results.
  Interventions: Behavioral: Video recording for behaviors

INTERVENTIONS:
Behavioral: Video recording for behaviors — A domenstic apparatus, scenario, and procedure is applied to record all the behavioral phenotypes.
  For each standardized procedure, the guardian sits in the chair, holding the infant facing the mobile phone screen. Each infant is given a few minutes to adapt to the surroundings and to be calm before recording. No hints or simulations are permitted during the entire process. The recording process lasted for about 3 minutes to ensure that behavioral phenotypes could be completely recorded.

SUMMARY:
An individual senses the world and reflects feedbacks via independent behaviors. Such precise collaboration of the sensory and behavioral systems is fundamental to survival and evolution. When a sensory modality is altered, the behavioral system has the potential to fit in a substitute modality. However, the specific dynamics of human behaviors in response to sensory loss remain largely unknown due to the paucities of representative situations and large-scale samples.

Here, the investigators focused on thousands of human infants who suffered varying degrees of visual stimuli deficiency in early stages, while their behavioral systems remained sensitive and thus retained high behavioral plasticity. Having access to this unique population provides an unprecedented opportunity to investigate the effect of diverse visual conditions on the behavioral system and develop a domestic apparatus for screening visual impariment of infants.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 4 years of age

Exclusion Criteria:

* Any brain and mental illnesses, or other known illnesses that may affect the behavioral patterns

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators focused on thousands of human infants who suffered varying degrees of visual stimuli deficiency in early stages, while their behavioral systems remained sensitive and thus retained high behavioral plasticity. Having access to this unique population provides an unprecedented opportunity to investigate the effect of diverse visual conditions on the behavioral system.
Sampling Method: Non-Probability Sample
Enrollment: 3652 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The AUC of model based on analyzing the behavioral dynamics | baseline
  Normal or abnormal behavioral dynamics of infants are recorded by mobile phones. Five experienced ophthalmologists identify the occurence of abnormal behaviors independently, and 2 professors with over 10 years of experience in pediatric ophthalmology department are consulted in cases of disagreement. The AUC of model based on analyzing the behavioral dynamics will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China